CLINICAL TRIAL: NCT06276374
Title: Clinical Trial to Obtain the Highest Efficacy of Dual Antiplatelet Therapy After Carotid Artery Stenting in High Bleeding Risk Patients
Brief Title: Highest Efficacy of Dual Antiplatelet Therapy After Carotid Artery Stenting in High Bleeding Risk Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Woo-Keun Seo (Other)
Responsible Party: Sponsor-Investigator, Woo-Keun Seo, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2023-12-107
Record Dates: First submitted 2024-02-13; First posted 2024-02-26 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Carotid Artery Diseases
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single antiplatelet therapy (SAPT) group with aspirin or clopidogrel (Experimental): 1 month of dual antiplatelet therapy(100mg aspirin q.d. and 75mg clopidogrel q.d.)→ Randomization → 11 months of single antiplatelet therapy (100mg aspirin q.d. or 75mg clopidogrel q.d.)
  Interventions: Drug: Patients who are scheduled to undergo carotid artery stenting
- Dual antiplatelet therapy (DAPT) with aspirin and clopidogrel (Active Comparator): 1 month of dual antiplatelet therapy(100mg aspirin q.d. and 75mg clopidogrel q.d.) → Randomization → 11 months of dual antiplatelet therapy (100mg aspirin q.d. and 75mg clopidogrel q.d.)
  Interventions: Drug: Patients who are scheduled to undergo carotid artery stenting

INTERVENTIONS:
Drug: Patients who are scheduled to undergo carotid artery stenting — * Arm A : Single antiplatelet therapy (SAPT) with aspirin or clopidogrel
    - 1 month of dual antiplatelet therapy(100mg aspirin q.d. and 75mg clopidogrel q.d.)→ Randomization → 11 months of single antiplatelet therapy (100mg aspirin q.d. or 75mg clopidogrel q.d.)
  * Arm B : Dual antiplatelet therapy (DAPT) with aspirin and clopidogrel - 1 month of dual antiplatelet therapy(100mg aspirin q.d. and 75mg clopidogrel q.d.) → Randomization → 11 months of dual antiplatelet therapy (100mg aspirin q.d. and 75mg clopidogrel q.d.)
  Other Names: Aspirin and,or Clopidogrel

SUMMARY:
To compare the safety of dual antiplatelet therapy with aspirin and clopidogrel and single antiplatelet therapy administered from 30 days to 12 months following carotid artery stenting on clinically significant bleeding and its prevention effects on net clinical events including combined cardiovascular and cerebrovascular accidents and major bleeding events in patients with carotid artery disease who are at high bleeding risk.

DETAILED DESCRIPTION:
* Arm A : Single antiplatelet therapy (SAPT) group

  - 1 month of dual antiplatelet therapy(100mg aspirin q.d. and 75mg clopidogrel q.d.) followed by 11 months of single antiplatelet therapy (100mg aspirin q.d. or 75mg clopidogrel q.d.)
* Arm B : Dual antiplatelet therapy (DAPT) with aspirin and clopidogrel - 1 month of dual antiplatelet therapy(100mg aspirin q.d. and 75mg clopidogrel q.d.) followed by 11 months of dual antiplatelet therapy (100mg aspirin q.d. and 75mg clopidogrel q.d.)

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥19 years
2. Symptomatic patients with carotid artery stenosis* greater than 50% and asymptomatic patients with carotid artery stenosis* greater than 70% who are scheduled to undergo or who have undergone carotid artery stenting
3. High bleeding risk is defined as a Bleeding Academic Research Consortium type 3 or 5 bleeding risk of ≥4% at 1 year or a risk of an intracranial hemorrhage (ICH) of ≥1% at 1 year, Patients who meet at least one of the criteria for high bleeding risk** below

   * The degree of stenosis is determined using the method performed in the North American Symptomatic Carotid Endarterectomy Trial.

     * Criteria for high bleeding risk (≥ 1)

       * Incidence of non-access site bleeding within 12 months prior to stenting (gastrointestinal tract or hematuria)
       * Presence of BARC type 3 or 5 bleeding regardless of the onset time, but the cause has not been completely cured.
       * Adults aged ≥75 years
       * Thrombocytopenia < 100,000/mm3 (based on the screening test)
       * Blood clotting disorders that increase bleeding (Von Willebrand disease, factor VII, VIII, IX, and XI deficiency)
       * Patients with anemia defined as hemoglobin <12g/dL in men and <11g/dL in women or patients who donated blood within 4 weeks (based on the screening test)
       * Patients received steroids or NSAIDs for ≥4 weeks
       * Patients with active malignancy (except for nonmelanoma skin cancer)
       * Renal disease (dialysis, transplantation, Estimated Glomerular Filtration Rate < 60ml/min per 1.73m2)
       * Liver disease (cirrhosis with portal hypertension)
       * Cerebral microbleeds ≥ 5
       * Stroke or transient ischemic attacks within 6 months or Transient amaurosis fugax
       * Incidence of nontraumatic intracerebral hemorrhage regardless of duration or incidence of traumatic intracerebral hemorrhage within 12 months

Exclusion Criteria:

1. Incidence of net clinical events, including cardiovascular and cerebrovascular accidents or major bleeding events, within 30 days following carotid artery stenting
2. Discontinuation of dual antiplatelet therapy within 30 days after carotid stent implantation (However, use of a single antiplatelet therapy within 7 days due to acute infection and trauma is allowed, but dual antiplatelet therapy must be administered at 28 to 30 days after carotid stent implantation)
3. Coronary artery stenting or other vascular stenting or vascular recanalization within 1 year (Revascularization surgery that requires CABG(Coronary Artery Bypass Graft) and other dual antiplatelet therapy)
4. Aspirin or clopidogrel hypersensitivity
5. Pregnant or breastfeeding women (Women of childbearing need to check for pregnancy using urine or blood tests before enrollment, and use appropriate contraception methods during the clinical trial period)
6. Patients requiring anticoagulation for ≥12 months
7. Patients requiring administration of other antiplatelet therapies
8. Patients who are participating in another intervention clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1556 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinically significant bleeding | From 30 days after carotid artery stenting until 12 months
  Bleeding Academic Research Consortium type 2, 3, or 5

SECONDARY OUTCOMES:
Combined cardiovascular and cerebrovascular accidents | From 30 days after carotid artery stenting until 12 months
  Combined outcome of nonfatal stroke, nonfatal myocardial infarction, death due to cardio- and cerebrovascular diseases, and major bleeding events

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No